CLINICAL TRIAL: NCT03209180
Title: Assessment of Clinical Effect and Treatment Quality of Rapid Release Carvedilol Versus SLOW Release Carvedilol-SR in HEART FAILURE Patient (SLOW-HF): A Prospective Randomized, Open-label, Multicenter Study
Brief Title: Immediate Release Versus Slow Release Carvedilol in Heart Failure
Acronym: SLOW-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, MD, PhD, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVDSR
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; Carvedilol; Slow Release; NT-proBNP

STUDY DESIGN:
Intervention Model Description: PROBE and NON-INFERIORITY DESIGN for Slow Release CarVeDilol-SR to Rapid Release Carvedilol-IR
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol IR (Immediate Release) (Active Comparator): Carvedilol IR 3.125mg, 6.25mg, 12.5mg, 25mg twice daily p.o. for 6 months
  Interventions: Drug: Carvedilol IR (Immediate Release)
- CarVeDilol-SR (Slow Release) (Experimental): CarVeDilol-SR 8mg, 16mg, 32mg, 64mg once daily p.o. for 6 months
  Interventions: Drug: CarVeDilol-SR (Slow Release)

INTERVENTIONS:
Drug: CarVeDilol-SR (Slow Release) — patients will receive slow-release carvedilol (SR) once daily
  Arms: CarVeDilol-SR (Slow Release)
Drug: Carvedilol IR (Immediate Release) — patients will receive immediate release carvedilol (IR) twice daily
  Arms: Carvedilol IR (Immediate Release)

SUMMARY:
Assessment of clinical effect and treatment quality of immediate release carvedilol (IR) versus slow release carvedilol (SR) in patients with HFrEF

DETAILED DESCRIPTION:
The SLOW-HF trial is a phase 4, randomized, open label, multicenter study to evaluate the therapeutic efficacy of carvedilol-SR compared to carvedilol-IR in patients with heart failure with reduced ejection fraction. Patients with stable HFrEF will be randomly assigned (1:1) to carvedilol SR group (160 patients) and carvedilol IR group (160 patients).

After randomization, patients will be followed for 6 months. The primary endpoint is the change in NT-proBNP level from baseline to the study end. The secondary endpoints include the frequency of NT-proBNP increment >10% from baseline, composite of all-cause mortality and readmission, mortality rate, readmission rate, changes in blood pressure, quality of life, and drug compliance.

ELIGIBILITY:
Inclusion criteria:

1. At least or more than 20-years-old male and female
2. Confirmed left ventricular ejection fraction ≤40% by echocardiography within pre-analytical 6 months
3. NT-proBNP level ≥ 125 pg/ml or BNP level ≥ 35 pg/ml within pre-analytical 3 months
4. Clinically stable patient without evidence of congestion or extracellular fluid retention; those could be candidate of β-blockers
5. Patients providing written informed consent

Exclusion Criteria:

1. Systolic blood pressure at sitting position < 90mmHg or resting heart rate < 50 /min at screening
2. Patient has a contraindication to β-blockers
3. Patient who are expected to take another β-blocker after randomization
4. Cardiovascular diseases

   * Ischemic heart disease (unstable angina, myocardial infarction) within 1 month
   * Hypertrophic cardiomyopathy
   * Cor pulmonale
   * Hemodynamically significant stenosis of aorta, aortic valve, or mitral valve
   * any acute myocardial infarction with complication
5. Severe cerebrovascular accident (for example, ischemic stroke or cerebral hemorrhage) pre-analytical within 6 months
6. Glottis edema, allergic rhinitis, respiratory diseases with bronchospasm such as asthma and chronic obstructive lung disease
7. Peripheral vascular disease (for example, Raynaud syndrome, intermittent claudication)
8. Patients who need vasopressor due to prominent volume retention/overload
9. Moderate to Severe retinopathy (for example, retinal hemorrhage, visual disturbance, retinal microaneurysm within 6 months)
10. Impaired renal function (Serum creatinine ≥ 2.5 mg/dL) or hepatic function (AST or ALT ≥ 3 x ULM)
11. Patients in clinical status that can significantly influence on absorption, distribution, metabolism, and secretion of drugs for clinical trial

    * history of major gastrointestinal surgery, such as gastrectomy or gastric bypass surgery
    * inflammatory bowel disease within 12 months
    * current gastric ulcer, pancreatic function abnormality including pancreatitis, gastrointestinal/rectal bleeding which demand treatment
    * current urologic stenosis or obstruction which demand treatment
12. Confirmed or suspected drug/alcohol abuse within 6 months
13. Pregnant or lactating women, suspected pregnant women or lactating women
14. Chronic inflammatory diseases which demand anti-inflammatory treatment
15. Hypersensitivity to carvedilol
16. Malignant disease including lymphoma and leukemia within 5 years
17. Patients who were prescribed other medication for any clinical trials pre-analytical within 28 days
18. Patients who are predicted to have prolonged hospital days due to other medical problems other than chronic heart failure (for example, femur neck fracture)
19. Patients who are considered as inappropriate to participate in the clinical trial by testers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-06-25 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | 6 months
  Change of NT-proBNP from baseline to 6 months after randomization

SECONDARY OUTCOMES:
All-cause Death | 6 months
  Difference in all-cause deaths between the groups during clinical follow-up
Hospitalization | 6 months
  Difference in hospitalization for heart failure between the groups during clinical follow-up
Blood Pressure | 6 months
  Difference in blood pressure change between the groups during clinical follow-up
Dyspnea | 6 months
  Differences in dyspnea measured with visual analogue scale between the groups during clinical follow-up
Drug compliance | 6 months
  Differences in drug compliance measured with 'pill-count' between the groups during clinical follow-up

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Sejong Hospital, Gyeonggi-do, Bucheon
  - Gangdong Sacred Heart Hospital, Seoul, Gangdong
  - Korea Univ. Guro Hospital, Seoul, Guro
  - Samsung Medical Center, Seoul, Il-won
  - Seoul Medical Center, Seoul, Jungnang
  - Korea Univ. Anam Hospital, Seoul, Seongbuk
  - Asan Medical Center, Seoul, Songpa
  - Ajou Univ. Medical Center, Suwon, Yeong-tong
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Park CS, Park JJ, Lee HY, Kang SM, Yoo BS, Jeon ES, Hong SK, Shin JH, Kim MA, Park DG, Kim EJ, Hong SJ, Kim SY, Kim JJ, Choi DJ. Clinical Characteristics and Outcome of Immediate-Release Versus SLOW-Release Carvedilol in Heart Failure Patient (SLOW-HF): a Prospective Randomized, Open-Label, Multicenter Study. Cardiovasc Drugs Ther. 2023 Jun;37(3):529-537. doi: 10.1007/s10557-021-07238-3. Epub 2022 Jan 23. PMID 35066737
- [Derived] Choi DJ, Park CS, Park JJ, Lee HY, Kang SM, Yoo BS, Jeon ES, Hong SK, Shin JH, Kim MA, Park DG, Kim EJ, Hong SJ, Kim SY, Kim JJ. Assessment of clinical effect and treatment quality of immediate-release carvedilol-IR versus SLOW release carvedilol-SR in Heart Failure patients (SLOW-HF): study protocol for a randomized controlled trial. Trials. 2018 Feb 13;19(1):103. doi: 10.1186/s13063-018-2470-5. PMID 29433525